CLINICAL TRIAL: NCT02604225
Title: A Phase 3 Double-blind Placebo-controlled Randomized Trial of Methoxyflurane With Periprostatic Local Anaesthesia to Reduce the Discomfort of Transrectal Ultrasound-guided Prostate Biopsy
Brief Title: Trial of Methoxyflurane With Periprostatic Local Anaesthesia to Reduce the Discomfort of TRUS B
Acronym: TRUSB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sydney (Other)
Collaborators: Australian and New Zealand Urogenital and Prostate Cancer Trials Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANZUP 1501; ACTRN12615001105538 (Registry Identifier: ANZCTR)
Record Dates: First submitted 2015-11-09; First posted 2015-11-13 (Estimated); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Cancer
Keywords: Anaethesiology
MeSH Terms: conditions — Neoplasms | interventions — Methoxyflurane; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Penthrox (Experimental): Methoxyflurane
  Interventions: Drug: Methoxyflurane
- Placebo (Placebo Comparator): Saline 0.9%
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methoxyflurane — Participants randomised to the experimental arm will inhale methoxyflurane administered through the Penthrox® inhaler starting approximately one minute before insertion of the rectal probe.
  Other Names: Penthrox®
  Arms: Penthrox
Drug: Placebo — Participants randomised to the control arm will inhale 0.9% saline administered through the Penthrox® inhaler starting approximately one minute before insertion of the rectal probe.
  Other Names: Saline 0.9%
  Arms: Placebo

SUMMARY:
A phase 3 double-blind placebo-controlled randomized trial of methoxyflurane with periprostatic local anaesthesia to reduce the discomfort of transrectal ultrasound-guided prostate biopsy (Pain-Free TRUS B).

DETAILED DESCRIPTION:
Background Transrectal ultrasound-guided (TRUS) prostate biopsy is associated with significant discomfort, despite the use of periprostatic infiltration of local anaesthetic (PILA).

General aim To determine the efficacy and safety of inhaled methoxyflurane plus PILA versus PILA alone in men undergoing TRUS biopsy of the prostate.

Objectives (endpoints)

To determine the effects of inhaled methoxyflurane on:

Primary

1. Pain-rated by participants 15 minutes after biopsy.

   Secondary
2. Other aspects of the biopsy experience rated by participants 15 minutes and 7-35 days after the biopsy
3. Willingness to undergo a biopsy in the future
4. Urologist's ratings of the participant's biopsy experience (study specific questionnaire completed after the biopsy)
5. Biopsy completion (80% or more of the planned number of biopsies being taken)
6. Frequency of specified adverse events (CTC AE v4.03 and Clavien-Dindo Classification).
7. Frequency of hospitalisation

Design Multi-centre, placebo-controlled, double-blinded, centrally randomised (1:1), stratified, phase 3 trial.

Target population Men scheduled to undergo their first TRUS biopsy of the prostate for a raised PSA or abnormal digital rectal examination (DRE).

Study treatments

Participants randomised to inhaled:

Methoxyflurane (Penthrox®, experimental group). OR Placebo (0.9% saline, control group

All participants are subsequently treated with PILA (2% lignocaine), injected into and around the prostate about 5 minutes before the biopsy.

Assessments Participants will be assessed at time of scheduling of the TRUS prostate biopsy (up to 84 days prior to randomisation), on the day of biopsy, and at the post biopsy clinic (7-35 days after the biopsy). Assessments comprise of medical history and standard blood tests at baseline, patient questionnaire on the day of biopsy and post(7-35 days) biopsy and safety assessments on the day of biopsy and post (7--35 days) biopsy.

Statistical considerations 420 participants provides over 85% power at the two-sided 5% level of significance to detect a 0.80 point difference in mean pain scores (on scale from 0-10) assuming a standard deviation of 2.5 whilst allowing for missing data. A 0.80 point shift in mean pain scores should correspond to a reduction of more than 1/3 in the proportion of men reporting troublesome levels of pain.

ELIGIBILITY:
Inclusion Criteria:

1. Males older than 18 years scheduled to undergo a TRUS biopsy of the prostate.
2. Adequate liver function: ALT, AST, or bilirubin ≤ 2 x ULN
3. Adequate renal function: serum eGFR> 30 ml/min/1.73m2
4. Willing and able to complete questionnaires in English
5. Willing and able to undergo TRUS biopsy within 7 days of randomisation
6. Willing and able to comply with all study requirements, including treatment, timing and/or nature of required assessments
7. Signed, written informed consent

Exclusion Criteria:

1. Previous TRUS biopsy of the prostate
2. Personal or family history of malignant hyperthermia
3. History of significant liver disease
4. Hypersensitivity to fluorinated anaesthetics or other inhalational anaesthetics
5. Concurrent use of barbiturates or tetracycline antibiotics
6. Concurrent illness that may jeopardise the ability of the patient to undergo the procedures outlined in this protocol with reasonable safety
7. Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule, including alcohol dependence or drug abuse.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2015-12; Primary Completion 2019-12-05 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Pain rated by participants will be self-rated using a numeric rating scale with verbal anchors from 0 (no trouble at all) to 10 (worst I can imagine). | Pain will be assessed at 15 minutes after the TRUS biopsy

SECONDARY OUTCOMES:
Other aspects of the biopsy experience rated by participants on the Patient's Experience of TRUS biopsy questionnaire. | Rated at 15 minutes after the biopsy
Other aspects of the biopsy experience rated by participants on the Patient's Experience of TRUS biopsy questionnaire. | Rated at 7-35 days after the biopsy
Willingness to undergo a biopsy in the future assessed by a questionnaire designed specifically for this study. | Rated at 15 minutes and 7-35 days after the biopsy
Urologist's ratings of the participant's biopsy experience, assessed by a questionnaire | On the same day as the TRUS biopsy
Biopsy completion rate. | Recorded on day of TRUS biopsy.
Frequency of specified adverse events. | Adverse events will be recorded after the TRUS biopsy (before the participant leaves the clinic), and 7-35 days after the biopsy.
Frequency of hospitalisation by reviewing hospital records. | Details will be recorded for each emergency department visit and each non-elective hospital admission that occurs within 30 days of the TRUS biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Grummet, Study Chair — Principal Investigator
Locations (7):
- Australia (6):
  - Concord Hospital, Concord, New South Wales
  - Australian Clinical Trials, Wahroonga, New South Wales
  - Casey Hospital, Berwick, Victoria
  - The Alfred Hospital, Prahran, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Westmead Hospital, Westmead
- Canterbury Urology Research Trust, Christchurch, New Zealand